CLINICAL TRIAL: NCT04267731
Title: Double Blinded, Randomized, Placebo Controlled Preliminary Pilot Exploratory Investigation Into the Effects of a Bifidobacterium Breve Extract, as VMK223, on Blood Inflammatory Markers, Gut Microbiota Composition and Tolerance in Healthy Adults Ages >50yrs Over a 3-week Period
Brief Title: Gut Health, Inflammation, Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vemico Ltd. (Industry)
Collaborators: University of Roehampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VMK1
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2022-04

CONDITIONS: Aging Well
Keywords: Gut microbiota; Postbiotics; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Cellulose; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo controlled, randomised dose response study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Cellulose 0.75g per day
  Interventions: Dietary Supplement: Cellulose
- Low dose (Experimental): 0.25g VMK223 per day
  Interventions: Dietary Supplement: VMK223
- Middle dose (Experimental): 0.5g VMK223 per day
  Interventions: Dietary Supplement: VMK223
- High dose (Experimental): 0.75g VMK223 per day
  Interventions: Dietary Supplement: VMK223

INTERVENTIONS:
Dietary Supplement: VMK223 — Heat killed and purified Bifidobacterium breve polysaccharide-based extract
  Other Names: Bifidobacterium breve extract/lysate
  Arms: High dose; Low dose; Middle dose
Dietary Supplement: Cellulose — Bulking agent in food production without probiotic properties
  Other Names: Cellulose microcrystalline
  Arms: Placebo

SUMMARY:
Pilot exploratory study on the effect of a Bifidobacterium breve extract, as VMK223, on plasma inflammatory markers, saliva hormones, gut microbiota and tolerance in females over 50years old. Participants are randomised in one of 4 arms: 0.25g/d VMK223, 0.5g/d VMK223, 0.75g/d VMK223, or placebo.

DETAILED DESCRIPTION:
The commensal bacteria colonising the gut and making up the microbiome perform a number of functions through their normal life cycle, which provide benefits to their human hosts in maintaining homeostasis. The relationship works both ways with the human host providing both nutrition and an environment for the bacteria to flourish.

Ageing is a natural and multifactorial phenomenon characterised by the accumulation of degenerative processes that are in turn underpinned by multiple alterations and damage within molecular pathways. The alterations and damage ultimately compromise cell and tissue functions. As such, ageing is the most profound risk factor for almost all non-communicable diseases. Amongst the key processes involved [in ageing], inflammation is of particular interest, because ageing is characterised by an increase in the concentration of a number of pro-inflammatory molecules in the circulation, a phenomenon that has been termed "inflammageing" and is a determinant of the speed of the ageing process and of lifespan.

Amongst the members of the human microbiome, Bifidobacterium spp. are resident microbiota members throughout the invesstigator's lifetime, with their levels across the life course aligning with key stages in immune maturation. Bifidobacteria influence this critical homeostatic development and programming by impacting on specific immune populations and signalling pathways associated with improved host well-being.

VMK223 is a heat treated Bifidobacterium breve extract, consisting of a low molecular weight storage polysaccharide that targets the reduction of NF-κB activation.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 50 years to 65 years
* Not dieting within the last month and not having lost >5% body weight in the previous year
* Not increased physical activity levels in the past 2-4 weeks or intending to modify them during the study
* Understands and is willing, able and likely to comply with all study procedures and restriction including being willing to follow the nutritional advice
* Able to eat most everyday foods
* Habitually consumes three standard meals a day

Exclusion Criteria:

* Significant health problems (e.g. hypercholesterolaemia, diabetes, GI disorders)
* Taking any medication or supplements known to affect immune system function within the past month and/or during the study
* Pregnant, planning to become pregnant or breastfeeding
* History of anaphylaxis to food
* Known allergies or intolerance to foods and/or to the study materials (or closely related compounds) or any of their stated ingredients
* Volunteers self-reporting currently dieting or having lost >5% body weight in the previous year
* Participants with abnormal eating behaviour
* Participation in another experimental study or receipt of an investigational drug/product within 30 days of the screening visit
* Volunteers who have significantly changed their physical activity in the past 2-4 weeks or who intend to change them during the study
* Participants receiving systemic or local treatment likely to interfere with the evaluation of the study parameters
* Participants on specific food avoidance diets
* Participants who work in appetite or feeding related areas

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Bowel Movements | 3 weeks
  self reported daily number of bowel movements
Stool form | 3 weeks
  self reported daily using the bristol 7-point scale (1:hard to 7:watery)
Flatulence | 3 weeks
  self reported daily using a 4-point scale (0: none, 3: severe)
Bloating | 3 weeks
  self reported daily using a 4-point scale (0: none, 3: severe)
Abdominal pain | 3 weeks
  self reported daily using a 4-point scale (0: none, 3: severe)

SECONDARY OUTCOMES:
C-Reactive protein | 3 weeks
  Plasma measurement
Interleukin-6 | 3 weeks
  Plasma measurement
Tumor Necrosis Factor alpha | 3 weeks
  Plasma measurement
Interleukin-10 | 3 weeks
  Plasma measurement
Interferon gamma | 3 weeks
  Plasma measurement
Human growth hormone | 3 weeks
  Plasma measurement
Cortisol | 3 weeks
  Saliva
Oestradiol | 3 weeks
  saliva
Oestriol | 3 weeks
  saliva
Progesterone | 3 weeks
  Saliva
Dehydroepiandrosterone | 3 weeks
  Saliva

OTHER OUTCOMES:
Positive and Negative Affect Schedule | 1 day
  Self reported positive/negative perception 5-point scale questionnaire. The positive affect score range is 10-50 and the negative affect score range is 10-50. Higher scores represent higher effect.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Costabile, Principal Investigator — University of Roehampton
Locations (1):
- University of Roehampton, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified participants data for all outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months after study completion
Access Criteria: Based on a data sharing agreement, a review panel will decide on all data sharing request